CLINICAL TRIAL: NCT03977805
Title: Metabolism and Disposition of [14C] Herombopag in Chinese Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HR-TPO-Ih
Record Dates: First submitted 2019-05-05; First posted 2019-06-06 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hetrombopag Olamine (Experimental): Hetrombopag Olamine (5 mg, 100 uCi)
  Interventions: Drug: Hetrombopag Olamine

INTERVENTIONS:
Drug: Hetrombopag Olamine — a single oral taking

SUMMARY:
This study is a single-center, open-label, single-dose design. It is planning to enroll six Chinese healthy adult male subjects. The metabolism and disposition of Herombopag, will be studied in these subjects after a single oral administration of a solution dose of [14C] Herombopag (5 mg, 100 uCi).

DETAILED DESCRIPTION:
The metabolism and disposition of Herombopag, will be studied in six healthy men after a single oral administration of a solution dose of [14C]eltrombopag (5 mg,100 uCi).

The sutdy will investigate total radioactivity pharmacokinetics in whole blood and plasma 、quantitatively analyze the the total radioactivity in the excreta、evaluate the predominant route of elimination and indentify the Metabolite profiles in plasma 、urine and faces.

ELIGIBILITY:
Inclusion Criteria:

* Health male subjects, age between 18-45 years.
* BMI between 19 and 26 kg/m2 .
* Signed informed consent.

Exclusion Criteria:

* Abnormal results in physical examination、laboratory tests、X-ray、abdominal ultrasound、echocardiography have clinical significance.
* Abnormal platelet counts or platelet aggregation has clinical significance.
* Abnormal troponin examination has clinical significance.
* Abnormal ophthalmic examination has clinical significance.
* Hepatitis B surface antigen, hepatitis C antibody, syphilis antibody or HIV antibody is positive.
* Those who have a history of allergies to test drugs or similar drugs.
* Those who have undergone surgery within 6 months prior to the trial .
* Those who took any drug within 14 days before the test (including Chinese herbal medicine).
* Any drug that inhibits or induces liver drug metabolism within 30 days before the test.
* Subjects who have participated in other clinical trial within the 3 months prior to study entry.
* One or more non-pharmacological contraceptive measures cannot be used during the trial or it is planned to have birth within one year.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-05-25 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Total radioactivity pharmacokinetics in whole blood and plasma | From 1 hour before administration to 240 hours after administration
  plasma concentration of total radioactivity
total radioactivity in the excreta | From 24 hour before administration to 336 hours after administration
  Excretion of radioactivity in human urine and feces
the concentration of Hetrombopag in plasma | From 1 hour before administration to 240 hours after administration
  Area under the plasma concentration versus time curve (AUC)
individual metabolite profiles in plasma 、urine and faces | From 24 hour before administration to 336 hours after administration
  Using quantitative High Performance Liquid Chromatography-Mass Spectroscopic method to analyse individual percentage of metabolites.
mean metabolite profiles in plasma 、urine and faces | From 24 hour before administration to 336 hours after administration
  Using quantitative High Performance Liquid Chromatography-Mass Spectroscopic method to analyse mean percentage of metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, PhD, Principal Investigator — First Affiliated Hospital of Suzhou Medical College
Locations (1):
- The first affiliated hospital of Suzhou university, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No